CLINICAL TRIAL: NCT05698485
Title: The Effects of a 3-Part Skin Care Regimen on Facial Wrinkles and Biophysical Attributes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Arbonne (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARB_SKIN3
Record Dates: First submitted 2023-01-06; First posted 2023-01-26 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: Wrinkle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3 Step Skin Care Regimen (Experimental): 3 different skin care products will be applied to the face
  Interventions: Other: Cleansing Balm; Other: Facial Serum; Other: Moisturizer

INTERVENTIONS:
Other: Cleansing Balm — DermResults Cleansing Balm w/ Avocado Oil twice daily
Other: Facial Serum — DermResults Advanced Serum w/ Hyaluronic Acid twice daily
Other: Moisturizer — DermResults Advanced Moisturizer w/ Hyaluronic Acid twice daily

SUMMARY:
The purpose of this study is to analyze various cosmetic endpoints, subjective assessments, and skin parameters such as hydration, transepidermal water loss, fine lines, and wrinkles with the use of a 3-part skin care regimen.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between the ages of 35 years old and 65 years old.
* Must have facial fine lines and wrinkles.

Exclusion Criteria:

* Individuals who are pregnant or breastfeeding.
* Prisoners
* Adults unable to consent
* Individuals who have changed any of their hormonal based contraception within 1 months prior to joining the study.
* Subjects using any topical retinoid, bakuchiol, hyaluronic acid or benzoyl peroxide containing topical product within 2 weeks of starting study or any subject unwilling to refrain from washout prior to enrollment.
* Subjects with any cosmetic treatments in the past 6 months and who are unwilling to withhold facial cosmetic treatments during the study including botulinum toxin, injectable fillers, microdermabrasion, intense pulsed light (IPL), peels, laser treatments, acid treatments, tightening treatments, facial plastic surgery, or any other medical treatment administered by a physician or skin care professional which is designed to improve the appearance of facial skin.
* Current tobacco smoker or a tobacco smoking history of greater than 10 pack-years

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-24 (Actual); Study Completion 2023-12-16 (Estimated)

PRIMARY OUTCOMES:
Appearance of facial wrinkles | 8 weeks
  Change in wrinkle severity measured by photographic analysis (BTBP 3D Camera System)

SECONDARY OUTCOMES:
Skin hydration | 1 week
  Change in skin hydration by SkinMoistureMeterSC measurement
Skin hydration | 4 weeks
  Change in skin hydration by SkinMoistureMeterSC measurement
Skin hydration | 8 weeks
  Change in skin hydration by SkinMoistureMeterSC measurement
Transepidermal water loss | 1 week
  Change in transepidermal water loss measurement by Vapometer
Transepidermal water loss | 4 weeks
  Change in transepidermal water loss measurement by Vapometer
Transepidermal water loss | 8 weeks
  Change in transepidermal water loss measurement by Vapometer
Skin volume | 1 week
  Change in skin volume/plumpness by photographic image analysis (BTBP 3D Camera System)
Skin volume | 4 weeks
  Change in skin volume/plumpness by photographic image analysis (BTBP 3D Camera System)
Skin volume | 8 weeks
  Change in skin volume/plumpness by photographic image analysis (BTBP 3D Camera System)
Skin texture/roughness | 1 week
  Change in the appearance of photographic analysis of texture/roughness with BTBP 3D Camera System
Skin texture/roughness | 4 weeks
  Change in the appearance of photographic analysis of texture/roughness with BTBP 3D Camera System
Skin texture/roughness | 8 weeks
  Change in the appearance of photographic analysis of texture/roughness with BTBP 3D Camera System
Self-perception of skin parameters | 1 week
  Survey based self-assessment of facial fine lines and wrinkles, skin smoothness, skin firmness
Self-perception of skin parameters | 4 weeks
  Survey based self-assessment of facial fine lines and wrinkles, skin smoothness, skin firmness
Self-perception of skin parameters | 8 weeks
  Survey based self-assessment of facial fine lines and wrinkles, skin smoothness, skin firmness
Tolerability of products | 1 week
  Questionnaire based self-assessment about the tolerability of the topical skin products
Tolerability of products | 4 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin products
Tolerability of products | 8 weeks
  Questionnaire based self-assessment about the tolerability of the topical skin products
Appearance of facial wrinkles | 4 weeks
  Change in wrinkle severity measured by photographic analysis (BTBP 3D Camera System)

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No